CLINICAL TRIAL: NCT04657588
Title: Controlling Faecal Incontinence With a Novel Anal Device: a Cost-effectiveness Trial (CONFIDEnCE)
Brief Title: Controlling Faecal Incontinence With a Novel Anal Device: a Cost-effectiveness Trial
Acronym: CONFIDEnCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 75495
Record Dates: First submitted 2020-10-13; First posted 2020-12-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-08

CONDITIONS: Faecal Incontinence
Keywords: faecal incontinence; Anal device; Navina anal insert; Self-help instrument
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Intervention Model Description: multicenter randomized controlled open-label superiority trial with adaptive design in ambulatory patients with FI with two parallel treatment arms: anal inserts and care as usual (incontinence pads).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anal insert (Experimental): This group will be asked to use anal inserts to help manage their faecal incontinence during the treatment period
  Interventions: Device: Navina anal insert
- Care as usual (Sham Comparator): This group will be asked to continue with their care as usual (e.g. incontinence pads)
  Interventions: Other: Care as usual

INTERVENTIONS:
Device: Navina anal insert — The Navina anal device is a single-use, pre-lubricated, liquid-filled rectal insert with a plastic applicator. The insert is filled with liquid mineral oil. The primary advantage of this new instrument is the fact that the liquid-filled insert will move and adapt as the fluid is transferred throughout the device making it easy to insert/remove and comfortable to wear. The design is intended to adjust to the contours of the individual anatomy to prevent leakage.
  Other Names: anal plug
  Arms: Anal insert
Other: Care as usual — Care as usual means participants are to continue their usual treatment for FI, like they would if they would not have participated in this study.
  Other Names: Comparator
  Arms: Care as usual

SUMMARY:
The purpose of this study is to assess the cost-effectiveness and improvement in quality of life of using a novel anal insert (navina)

DETAILED DESCRIPTION:
After being informed about the study including the potential pros and cons, patients will be given a minimum of 7 days to think about whether they would like to participate in the study. If they would like to participate, and informed consent form will need to be signed, after which the patients will undergo a screening to ensure they meet the inclusion criteria. A 2 week run-in period will take place to let patients get used to filling in an electronic daily diary. Prior to this period, patients will be asked to fill out several questionnaires. After this period, randomisation into either (1) the anal insert group or (2) the care as usual group. Group 1 will then have an 'accommodation' week in which they can try out two different sizes of the anal insert to see which size they would prefer for the treatment period. The treatment period will consist of 8 weeks In which the (1) anal insert group is expected to use the anal inserts and the (2) care as usual group is asked to continue with their treatment as usual. During the treatment period, patients will fill out an electronic daily diary as well as weekly questionnaires.At the end of the 8 week treatment period, patients will fill out additional questionnaires. The follow-up consists of 4 weeks, after which patients will be asked again to fill out several questionnaires.

ELIGIBILITY:
Inclusion Criteria:

For run in period

* Patients with FI according to Rome IV criteria (i.e. recurrent uncontrolled passage of faecal matter for at least 3 months)
* Aged between 16-90 years

For randomisation and treatment period

* Patients with FI according to Rome IV criteria (i.e. recurrent uncontrolled passage of faecal matter for at least 3 months)
* Aged between 16-90 years
* patients who experience at least 1 episode of accidental bowel leakage during the 2 week run-in period will be eligible for randomisation.

Exclusion Criteria:

* Insufficient cognitive skills to fill in patient-reported questionnaires, inability to present to hospital for screening visit and inclusion, neurological/psychiatric or physical inability to comply with the study protocol (including diary assessments) at the investigator's discretion, or insufficient command of the Dutch language.
* Anatomic abnormalities: known communication between the anal and vaginal tracts, prior diagnosis of congenital anorectal malformations, previous rectal surgery, radiotherapy to a pelvic organ (uterus, prostate, rectum).
* Prior diagnosis of inflammatory bowel disease.
* Pregnancy or intention to become pregnant during the study period.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in FI severity | 8 weeks
  Measured using the St. Marks/vaizey incontinence score. This scale ranges from 0 (complete continence = best score) to 24 (complete incontinence= worst score). We are particularly interested in whether a clinically meaningful decrease of ≥3 points will occur in the intervention group compared to the control group.

SECONDARY OUTCOMES:
Cost effectiveness (direct medical costs) | 8 weeks
  Determined through the Medical consumption questionnaire (MCQ).
Cost effectiveness (Costs due to loss of productivity) | 8 weeks
  Determined through the Productivity Cost Questionnaire (PCQ).
Mental health (anxiety) | 8 weeks
  Measured through the Generalized anxiety disorder (GAD-7) questionnaire. This questionnaire contains 7 questions which can each be given a score of 0 to 3. A total score of 0= no anxiety (the best), a total score of 21= severe anxiety (the worst)
Mental health (depression) | 8 weeks
  Measured through the Patient health questionnaire 9 (PHQ-9).
Quality of life (QoL) (general QoL) | 8 weeks
  Measured through the 5 level EQ-5D questionnaire (EQ-5D-5L). This questionnaire contains 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) which can all individually be scored on a scale of 0 (best) to 5(worst). Additionally participants are asked to score their health for that day from a score of 0 (worst health you can imagine) to a score of 100 (best health you can imagine).
Quality of life (QoL) (disease specific QoL) | 8 weeks
  Measured through the Faecal incontinence Quality of life scale (FIQL). This questionnaire contains 24 items which can be scored from 1( worst) to 4,5 or 6 (best) depending on the item. Patients can score a minimum of 29 points (worst QoL) to a maximum of 119 points (best QoL).
Adherence to therapy | 8 weeks
  Checking whether patients in the anal insert group (intervention) decided to use the anal inserts or not
Wellbeing | 8 weeks
  Measured through the ICEpop CAPability measure for adults (ICE-CAP-A) questionnaire. To measure wellbeing in terms of capabilities like attachment; security (thinking about the future without concern); role (doing things that make you feel valued); enjoyment and pleasure; control (independence). Each of the 5 items can be given a score of 1 (worst) to 4 (best).
Frequency and severity of adverse events | 8 weeks
  Any adverse events possibly related to the anal insert will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No